CLINICAL TRIAL: NCT02909218
Title: MaxART: Early Access to ART for All in Swaziland
Acronym: MaxART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinton Health Access Initiative Inc. (Other)
Collaborators: Ministry of Health, Swaziland (Other Government); STOP AIDS NOW! (SAN!) (Unknown); Swaziland National Network of People Living with HIV/AIDS (SWANNEPHA) (Unknown); Southern African AIDS Information Dissemination Service (SAfAIDS) (Unknown); Southern African Centre for Epidemiological Modelling and Analyses (SACEMA) (Unknown); University of Amsterdam (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MaxART
Record Dates: First submitted 2016-07-10; First posted 2016-09-21 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS, Swaziland
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- National HIV Treatment Guidelines (No Intervention): HIV-positive individuals are offered ART per Swaziland's national treatment guidelines
- Early Access to ART for All (Experimental): HIV-positive individuals are initiated on ART regardless of client's immunological and clinical staging
  Interventions: Other: Early Access to ART for All

INTERVENTIONS:
Other: Early Access to ART for All — All HIV-positive individuals will be initiated on Swaziland's recommended first-line ART regimen, unless contraindicated when recommended alternate regimens will be used per national guidelines.
  Arms: Early Access to ART for All

SUMMARY:
The purpose of this study is to evaluate the feasibility, acceptability, clinical outcomes, affordability, and scalability of offering early antiretroviral treatment to all HIV-positive individuals in Swaziland's government-managed health system.

DETAILED DESCRIPTION:
The clinical evidence in support of offering antiretroviral treatment (ART) for all HIV-positive individuals to improve patient health outcomes and reduce HIV incidence is building, and the resource-limited countries where this approach could have the biggest impact want to evaluate if this is a feasible and effective intervention to turn the course of their HIV epidemics. The MaxART Early Access to ART for All (EAAA) implementation study was designed to determine the feasibility, acceptability, clinical outcomes, affordability, and scalability of offering early antiretroviral treatment to all HIV-positive individuals in Swaziland's government-managed health system.

This is a 3-year randomized stepped wedge design with open enrollment for all adults 18 years and older across 14 rural health facilities in Swaziland's Hhohho Region. Primary endpoints are retention and viral suppression. Secondary endpoints include ART initiation, adherence, drug resistance, tuberculosis, HIV disease progression, and cost per patient per year.

Sites are grouped to transition two at a time from the control (standard of care) to intervention (EAAA) stage at each 4-month step. This balanced design will result in approximately one half of the observations being under an intervention clinic, and the other half under control.

Power calculations were conservatively based on the estimated number of individuals expected to enroll in the study comparing the first 12-month measure of retention and 6-month of viral suppression on ART of those entering clinics during their control stage versus those that will be entering a clinic during intervention period.

A strategic mix of multidisciplinary research methodologies will be applied to meet the study aim, including implementation science, social science research, economic evaluations, and HIV incidence modeling.

ELIGIBILITY:
Inclusion Criteria:

* All ART-naive HIV-positive individuals who are 18 years of age or older - excluding pregnant or breastfeeding women - who attend the health facilities included in the study will be asked for their consent to enroll in the study.

Exclusion Criteria:

* All HIV-positive individuals who < 18 years of age or older and pregnant or breastfeeding women.
* All HIV-positive individuals who did not consent to participate or who have already been initiated on ART.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3485 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Retention | 12 months
  Proportion of individuals retained in care or on ART at 12 months
Viral suppression | 6 months
  Proportion of individuals whose viral load is below 1,000 copies/ml (virally suppressed) after 6 months on ART

SECONDARY OUTCOMES:
12-month mortality rate | 12 months
  mortality rate among clients newly enrolled in or returning to facilities during the standard of care phase is equal to 12-month mortality rate among clients newly enrolled in or returning to facilities during early ART phase
Visit adherence among those initiated on ART | 36 months
  Proportion of missed visits as a number of scheduled appointments among ART-ineligible clients by end of follow-up
Drug resistance | 36 months
  Proportion of drug resistance among ART-ineligible clients with two virological failures who have received genotype resistance testing
Tuberculosis | 36 months
  Proportion of HIV-positive individuals diagnosed with new tuberculosis following enrollment (recurrent and newly incident).
ART uptake among those who are eligible | 3 months
  Proportion of HIV-positive individuals who are eligible for initiation who are successfully initiated to ART within 1 and 3 months of becoming eligible
Cost per patient per year | 12 months
  Bottom-up and top-town costing of the patient lifetime cost to test, treat, link, and retain individuals on ART
HIV infection | 36 months
  Mathematical modeling to estimate the number of new adult HIV infections using empirical data from the primary endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Velephi Okello, MD, Principal Investigator — Ministry of Health, Swaziland
Locations (1):
- Swaziland Ministry of Health, Mbabane, Eswatini

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Briggs J, Teyssier N, Nankabirwa JI, Rek J, Jagannathan P, Arinaitwe E, Bousema T, Drakeley C, Murray M, Crawford E, Hathaway N, Staedke SG, Smith D, Rosenthal PJ, Kamya M, Dorsey G, Rodriguez-Barraquer I, Greenhouse B. Sex-based differences in clearance of chronic Plasmodium falciparum infection. Elife. 2020 Oct 27;9:e59872. doi: 10.7554/eLife.59872. PMID 33107430
- [Derived] Mobegi FM, Leong LE, Thompson F, Taylor SM, Harriss LR, Choo JM, Taylor SL, Wesselingh SL, McDermott R, Ivey KL, Rogers GB. Intestinal microbiology shapes population health impacts of diet and lifestyle risk exposures in Torres Strait Islander communities. Elife. 2020 Oct 19;9:e58407. doi: 10.7554/eLife.58407. PMID 33074097
- [Derived] Steinert JI, Khan S, Mlambo K, Walsh FJ, Mafara E, Lejeune C, Wong C, Hettema A, Ogbuoji O, Vollmer S, De Neve JW, Mazibuko S, Okello V, Barnighausen T, Geldsetzer P. A stepped-wedge randomised trial on the impact of early ART initiation on HIV-patients' economic outcomes in Eswatini. Elife. 2020 Aug 24;9:e58487. doi: 10.7554/eLife.58487. PMID 32831169
- [Derived] Walsh FJ, Barnighausen T, Delva W, Fleming Y, Khumalo G, Lejeune CL, Mazibuko S, Mlambo CK, Reis R, Spiegelman D, Zwane M, Okello V. Impact of early initiation versus national standard of care of antiretroviral therapy in Swaziland's public sector health system: study protocol for a stepped-wedge randomized trial. Trials. 2017 Aug 18;18(1):383. doi: 10.1186/s13063-017-2128-8. PMID 28821264